CLINICAL TRIAL: NCT05546957
Title: A Parallel Group Study in Healthy Participants to Quantify Subclinical Gastrointestinal Blood Loss Following Administration of Aspirin Alone or Aspirin in Combination With Rivaroxaban
Brief Title: Assess Gastrointestinal Blood Loss After Receiving Aspirin or Aspirin Plus Rivaroxaban in Healthy Adult Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R0000-HV-2229; 2022-002761-15 (EudraCT Number)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteer
Keywords: No gastrointestinal (GI) disease; No risk factors for bleeding; Direct oral anticoagulant (DOAC); Fecal occult blood testing (FOBT)
MeSH Terms: conditions — Disease | interventions — Aspirin; Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Aspirin QD (Experimental): Randomized 1:1:1
  Interventions: Drug: Aspirin
- Arm 2: Aspirin QD + rivaroxaban BID (Experimental): Randomized 1:1:1
  Interventions: Drug: Aspirin; Drug: rivaroxaban low dose
- Arm 3: Aspirin QD + rivaroxaban QD (Experimental): Randomized 1:1:1
  Interventions: Drug: Aspirin; Drug: rivaroxaban high dose

INTERVENTIONS:
Drug: Aspirin — Administered orally once per day (QD)
Drug: rivaroxaban low dose — Administered orally twice per day (BID)
  Arms: Arm 2: Aspirin QD + rivaroxaban BID
Drug: rivaroxaban high dose — Administered orally QD
  Arms: Arm 3: Aspirin QD + rivaroxaban QD

SUMMARY:
The primary objective of the study is to determine whether aspirin alone or aspirin combined with various doses of rivaroxaban causes subclinical GI blood loss as determined by the HemoQuant assay.

The secondary objective of the study is to evaluate the safety and tolerability of aspirin alone or in combination with rivaroxaban to healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index between 18 and 32 kilograms per metered square (kg/m2), inclusive
2. Is judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and electrocardiograms (ECGs) performed during screening
3. Is in good health based on laboratory safety testing obtained at the screening visit
4. Willing and able to abstain from alcohol use for the duration of the study

Key Exclusion Criteria:

1. History of anemia, abnormal bleeding (including vaginal bleeding or excessive menstrual periods), previous diagnosis of bleeding diathesis, or blood clots as defined in the protocol
2. History, in the last year, of any bleeding GI lesions such as peptic ulcer, hemorrhoids or anal fissure, or a positive fecal occult blood test performed either during screening or on Day 1
3. Presence of irregular stool patterns, constipation, or frequent diarrhea that, in the opinion of the investigator, may interfere with stool collections required by the protocol
4. Inability to refrain during study period from activities with high risk of bleeding or trauma such as planned surgery, contact sports, etc.
5. Hemoglobin levels below the lower limit of normal as defined by local laboratory at screening; the lab may be repeated once if initially abnormal
6. PT and aPTT values above the upper limit of normal as defined by the local laboratory during screening; the lab may be repeated once if initially abnormal
7. Platelet count below the lower limit of normal as defined by the local laboratory during screening; the lab may be repeated once if initially abnormal
8. History of clinically significant respiratory, hepatic, renal, GI, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator that may confound the results of the study or poses an additional risk to the participant by study participation.

   History of any atherosclerotic cardiovascular disease
9. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
10. Has received a COVID-19 vaccination within 1 week of day 1 of the study or for which the planned COVID-19 vaccinations would not be completed 1 week prior to day 1 of the study.

NOTE: Other protocol defined inclusion / exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fecal hemoglobin content as measured by HemoQuant during the second week of exposure to study medication | Up to Week 4
  HemoQuant is a chemical laboratory test of fecal hemoglobin content.

SECONDARY OUTCOMES:
Number of bleeding events during the baseline period as compared to the treatment period | Up to week 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- LabCorp CRU, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/